CLINICAL TRIAL: NCT02225132
Title: Assessment of Computerized Algorithm-Based Hydroxyurea Dosing on Fetal Hemoglobin Response, Acute Complications, and Organ Function in Subjects With Sickle Cell Disease
Brief Title: Assessment of Algorithm-Based Hydroxyurea Dosing on Fetal Hemoglobin Response, Acute Complications, and Organ Function in People With Sickle Cell Disease
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 140172; 14-H-0172
Record Dates: First submitted 2014-08-23; First posted 2014-08-26 (Estimated); Results first posted 2019-08-06 (Actual); Last update posted 2019-08-06 (Actual); Status verified 2019-04-25

CONDITIONS: Sickle Cell Disease
Keywords: Hydroxyurea; Sickle Cell Disease; Fetal Hemoglobin Induction
MeSH Terms: conditions — Anemia, Sickle Cell | interventions — Hydroxyurea

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- 1 (Experimental): This is a one arm, open-label, non- randomized pilot study to evaluate the effect of algorithm- based HU dosing on the HbF response, the ability to titrate each patient to the MTD of HU, acute complications, and organ function in patients with HbSS.
  Interventions: Drug: Hydroxyurea

INTERVENTIONS:
Drug: Hydroxyurea — The precise mechanism by which hydroxyurea produces its cytotoxic and cytoreductive effects is not known. However, various studies support the hypothesis that hydroxyurea causes an immediate inhibition of DNA synthesis by acting as a ribonucleotide reductase inhibitor, without interfering with the synthesis of ribonucleic acid or of protein.
  The mechanisms by which DROXIA produces its beneficial effects in patients with sickle cell anemia (SCA) are uncertain. Known pharmacologic effects of DROXIA that may contribute to its beneficial effects include increasing hemoglobin F levels in RBCs, decreasing neutrophils, increasing the water content of RBCs, increasing deformability of sickled cells, and altering the adhesion of RBCs to endothelium.

SUMMARY:
Background:

- Sickle cell disease (SCD) is a blood disease. The drug hydroxyurea (HU) is approved to prevent pain crises in people with SCD. Researchers want to see how higher doses of HU affect the blood. This will help them learn about the right dosage of HU to give to people with SCD.

Objective:

- To improve hydroxyurea dosing in people with SCD.

Eligibility:

- People age 15 or older with homozygous SCD (HbSS).

Design:

* Participants will be screened with medical history, physical exam, medication review, and blood and urine tests.
* Participants will be in the study for about 15 months.
* First 3 months: monthly study visits with blood and urine tests.
* After 3 months: participants will take HU as a capsule by mouth. If you are already taking HU, your dose will be increased.
* Within a month of starting or increasing HU: participants will keep a daily pain diary for 2 weeks. They will have an echocardiogram (ultrasound) of the heart, a 6-minute walk test. They will complete a quality-of-life questionnaire.
* Participants will visit every month until they reach their highest tolerated dose of HU. They may need to come as often as every week sometimes to closely monitor their blood counts. Then they will alternate a phone call one month and a visit the next. At the visits, participants will bring their pill bottle, answer questions about side effects, and have blood tests.
* Every 2 months, participants will have a medical history, physical exam, and blood tests.
* Every 4 months, participants will have blood and urine tests. They will also complete another 2-week pain diary and quality-of-life questionnaire.
* About 12 months after starting or increasing HU, participants will have blood tests, an echocardiogram, and a 6-minute walk test.

DETAILED DESCRIPTION:
Sickle cell disease (SCD) is associated with significant morbidity and early mortality. Despite the discovery of the disease more than 100 years ago, only one drug, hydroxyurea (HU), has been FDA-approved. Hydroxyurea exerts its beneficial effects largely by inducing fetal hemoglobin (HbF) and thereby inhibiting red blood cell sickling. Hydroxyurea has been shown to decrease the frequency of acute complications such as painful crises and acute chest syndrome. However, previous studies are conflicting regarding whether HU improves survival; 2 long-term studies where HU was titrated to the maximum tolerated dose show that HU improves survival. However, multiple studies performed in the era post-FDA approval of HU show no change in median survival. We and others have found that patients with SCD who die prematurely have more evidence of renal, hepatic, and cardiopulmonary damage. Our work also suggests that HU treatment per se is not sufficient to improve survival and decrease organ damage in patients with homozygous SCD (HbSS). Instead, patients treated with the highest HU doses and who had the highest HbF levels appeared more likely to survive and had less evidence of organ damage over time. Hydroxyurea management can be intimidating; therefore, many adults with HbSS are either not treated with HU or are treated with doses below that which are FDA-approved. A HU dosing algorithm may simplify dosing such that not only are more patients treated with HU, but more may be titrated to the maximal tolerated dose which may be necessary to prevent organ damage and prolong survival. Further, myelosuppression beyond what has traditionally been recommended may further maximize HbF response. This protocol is a prospective pilot study which follows a 2 month run-in period. Hydroxyurea dosing will be based on a written algorithm which will be derived manually, and by a computer program which was developed at the NIH Clinical Center. Clinical, laboratory, and echocardiographic parameters will be monitored at baseline and after treatment to further study the effect of maximum HbF response on acute complications associated with HbSS and organ function.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Age greater than or equal to 15 years
  2. Homozygous sickle cell disease (HbSS)
  3. Patients with recent transfusion must have HbA <15% prior to enrollment
  4. ANC greater than or equal to 2,000/microL, platelets greater than or equal to150,000/microL, Hb > 5.4g/dL, and ARC greater than or equal to100,000/microL (unless the Hb is > 8g/dL) at baseline
  5. Patients on angiotensin-converting enzyme inhibitors and angiotensin receptor blockers should be on a stable dose for 2 weeks prior to initiating or adjusting HU

EXCLUSION CRITERIA:

1. Pregnant or lactating women or patients planning to get pregnant during the study period
2. Patients unwilling to use two forms of contraception throughout the period of HU administration
3. Patients receiving chronic transfusion therapy
4. Patients receiving a HU dose of greater than or equal to 20 mg/kg/day
5. Patients with history of allergy or intolerance to HU judged by the investigator to be prohibitive against restarting HU

6 Patients with end stage renal disease defined as GFR <10mL/min/1.73m(2)

7. Patients being treated with antiretroviral agents (such as didanosine and stavudine) because of a higher risk for potentially fatal pancreatitis, hepatic failure, hepatitis, and severe peripheral neuropathy when co-administered with hydroxyurea.

8. Participation on any other chronic investigative treatment studies

9. Unable to understand the investigational nature of the study or give informed consent.

Ages: 15 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2014-08-23; Primary Completion 2018-05-24 (Actual); Study Completion 2018-05-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Courtney D Fitzhugh, M.D., Principal Investigator — National Heart, Lung, and Blood Institute (NHLBI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2014-H-0172.html

RESULTS

PARTICIPANT FLOW:
Groups:
- Hydroxyurea: Hydroxyurea is given to the patients as per a dosing algorithm.
Period: Overall Study
Arm/Group | Hydroxyurea
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Hydroxyurea
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 10
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 10
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 10
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Fetal Hemoglobin Level
Description: Mean fetal hemoglobin calculated to indicate effectiveness of hydroxyurea dose
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | Hydroxyurea
Number analyzed (Participants) | 10
Percentage | 8.3 (5.9)

2. Primary Outcome: Fetal Hemoglobin Level
Description: Mean fetal hemoglobin calculated to indicate effectiveness of hydroxyurea dose
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | Hydroxyurea
Number analyzed (Participants) | 10
Percentage | 25.1 (6.2)

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | Hydroxyurea
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 3/10
Other Adverse Events (participants affected / at risk) | 10/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Hydroxyurea (N=10)
Acute chest syndrome (Blood and lymphatic system disorders) | 1
Sickle cell anaemia with crisis (Blood and lymphatic system disorders) | 2
Viral infection (Infections and infestations) | 1
Knee arthroplasty (Surgical and medical procedures) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Hydroxyurea (N=10)
Anaemia (Blood and lymphatic system disorders) | 2
Blood disorder (Blood and lymphatic system disorders) | 5
Lymph node pain (Blood and lymphatic system disorders) | 1
Dizziness (Cardiac disorders) | 2
Dyspnoea (Cardiac disorders) | 2
Oedema peripheral (Cardiac disorders) | 2
Vision blurred (Eye disorders) | 1
Vitreous floaters (Eye disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 3
Vomiting (Gastrointestinal disorders) | 2
Fatigue (General disorders) | 2
Influenza like illness (General disorders) | 1
Pain (General disorders) | 8
Pyrexia (General disorders) | 2
Bronchitis (Infections and infestations) | 1
Upper respiratory tract infection (Infections and infestations) | 1
Alanine aminotransferase increased (Investigations) | 2
Neutrophil count decreased (Investigations) | 7
Platelet count decreased (Investigations) | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Headache (Nervous system disorders) | 4
Insomnia (Nervous system disorders) | 1
Nervous system disorder (Nervous system disorders) | 1
Somnolence (Nervous system disorders) | 1
Chromaturia (Renal and urinary disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Dermatitis bullous (Skin and subcutaneous tissue disorders) | 1
Nail discolouration (Skin and subcutaneous tissue disorders) | 2
Pruritus (Skin and subcutaneous tissue disorders) | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 3
Skin disorder (Skin and subcutaneous tissue disorders) | 1
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 3
Embolism (Vascular disorders) | 1
Thrombophlebitis superficial (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-08-23): https://cdn.clinicaltrials.gov/large-docs/32/NCT02225132/Prot_SAP_000.pdf